CLINICAL TRIAL: NCT03556215
Title: Balloon Eustachian Tuboplasty in Treatment of Chronic Eustachian Tube Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: University Hospital Hradec Kralove (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-ENT-BET; MH CZ - DRO - FNOs/2016 (Other Grant/Funding Number: Ministry of Health of the Czech Republic)
Record Dates: First submitted 2018-05-20; First posted 2018-06-14 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Chronic Eustachian Tube Dysfunction; Chronic Recurrent Otitis Media; Effusion After Tympanostomy
Keywords: otitis media with effusion; balloon tuboplasty; Eustachian tube; Eustachian tube dysfunction
MeSH Terms: conditions — Otitis Media with Effusion | interventions — Middle Ear Ventilation

STUDY DESIGN:
Intervention Model Description: Interventional parallel randomized controlled prospective trial
Masking Description: No masking was used in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Effusion, Eustachian tube dilatation device and myringotomy (Experimental): Patients with chronic Eustachian tube dysfunction and recurrence of chronic otitis media with effusion after tympanostomy tube exclusion, intervention: balloon Eustachian tuboplasty, and myringotomy
  Interventions: Device: Eustachian tube dilatation device; Procedure: Myringotomy
- Effusion, Eustachian tube dilatation device (Experimental): Patients with chronic Eustachian tube dysfunction and recurrence of chronic otitis media with effusion after tympanostomy tube exclusion, intervention: balloon Eustachian tuboplasty only (no myringotomy)
  Interventions: Device: Eustachian tube dilatation device
- No effusion, Eustachian tube dilatation device (Experimental): Patients with chronic Eustachian tube dysfunction and airy middle ear (without otitis media with effusion), Eustachian tube dilatation device, no myringotomy
  Interventions: Device: Eustachian tube dilatation device

INTERVENTIONS:
Device: Eustachian tube dilatation device — Balloon Eustachian tuboplasty will be performed using a Eustachian tube dilatation device.
Procedure: Myringotomy — Myringotomy will be performed using a standard procedure.
  Arms: Effusion, Eustachian tube dilatation device and myringotomy

SUMMARY:
The prevalence of Eustachian tube (ET) dysfunction in adults reaches 1%. It causes a feeling of fullness in the ear, otalgia and hearing loss and can lead to recurrent acute otitis media, development of chronic otitis media with effusion and cholesteatoma. Endoscopic transnasal balloon ET dilatation is a novel surgical technique for ET dysfunction. The main goal is to restore ET function by dilation its cartilaginous part leading to better ventilation and drainage of the middle ear. However, its real effect in the treatment of particular subgroups of patients with ET dysfunction remains unknown. Patients are mostly evaluated as one group.

Adults with chronic ET dysfunction will be strictly divided into particular subgroups and included in the study. Subgroups will be compared in order to identify treatment effect in particular subgroups.

DETAILED DESCRIPTION:
The prevalence of Eustachian tube (ET) dysfunction in adults reaches 1%. It causes a feeling of fullness in the ear, otalgia and hearing loss and can lead to recurrent acute otitis media, development of chronic otitis media with effusion and cholesteatoma. Endoscopic transnasal balloon ET dilatation is a novel surgical technique for ET dysfunction. The main goal is to restore ET function by dilation its cartilaginous part leading to better ventilation and drainage of the middle ear. However, its real effect in the treatment of particular subgroups of patients with ET dysfunction remains unknown. Patients are mostly evaluated as one group.

Adults with chronic ET dysfunction will be strictly divided into particular subgroups and included in the study. The otomicro(endo)scopy, symptoms severity according to VAS (Visual Analogue Pain Scale), ETDQ-7 (Eustachian Tube Dysfunction Questionnaire) questionnaire, tympanometry, audiometry and the possibility of Valsalva and Toynbee maneuver will be used to evaluate the effect of balloon ET dilatation. Only patients with standard treatment failure will be included in the study. Tuboplasty with and without myringotomy will be performed (and compared) in patients with chronic otitis media with effusion. Subgroups will be compared in order to find patients who could profit from the treatments the most.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with chronic Eustachian tube dysfunction lasting more than 6 months, with or without recurrence of chronic otitis media with effusion after tympanostomy

Exclusion Criteria:

* anatomic obstruction in nasopharynx
* nasopharyngeal cancer
* head and neck cancer
* other middle ear surgery except for myringotomy or tympanostomy
* chronic suppurative otitis media
* patients who could not undergo general anesthesia
* patients who did not give consent to be included in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Otomicro(endo)scopy | 36 months
  Otomicro(endo)scopy will be used to assess the presence or absence of effusion.

SECONDARY OUTCOMES:
Symptoms severity according to Visual Analogue Scale | 36 months
  Symptoms severity will be assessed on Visual Analogue Scale (on the scale of 1-10). Visual Analogue Scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
ETDQ-7 questionnaire | 36 months
  The patients will be asked to fill-in the Eustachian Tube Dysfunction Questionnaire in order to assess the symptoms of Eustachian Tube Dysfunction (ETD). The ETDQ-7 is a valid and reliable symptom score for use in adult patients with ETD. The ETDQ-7 tool consists of seven items with a scale of graduated responses ranging from 1 to 7, with "1" corresponding to the absence of the suggested symptom and "7", to maximum symptom severity.
Tympanometry | 36 months
  Type of tympanometry curve (A, B, C) according to Joerger et al.
Audiometry | 36 months
  Hearing loss according to WHO classification (mild, moderate, severe).
Tubomanometry | 36 months
  Assessment of opening pressure in Eustachian tube in mmHg.
Possibility of Valsalva and Toynbee manoeuvre | 36 months
  The possibility or inability of Valsalva and Toynbee manoeuvre (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Komínek, prof.,MD,Ph.D.,MBA, Study Chair — University Hospital Ostrava; Martin Formánek, MD, Principal Investigator — University Hospital Ostrava
Locations (2):
- Czechia (2):
  - University Hospital Hradec Králové, Hradec Králové, Hradec Králové Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Swords C, Smith ME, Patel A, Norman G, Llewellyn A, Tysome JR. Balloon dilatation of the Eustachian tube for obstructive Eustachian tube dysfunction in adults. Cochrane Database Syst Rev. 2025 Feb 26;2(2):CD013429. doi: 10.1002/14651858.CD013429.pub2. PMID 40008607